CLINICAL TRIAL: NCT03827382
Title: Bicycle Exercise and Lifestyle Intervention in Newly Diagnosed Diabetes
Acronym: BELIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Olten (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01920
Record Dates: First submitted 2018-12-06; First posted 2019-02-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Life Style
Keywords: Life Style Intervention; Type 2 Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Patients with intensive Lifestyle intervention
  Interventions: Behavioral: Lifestyle Intervention
- Control (No Intervention): Patients with Standard Diabetes care

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Physical activity program: 3-5 aerobic training sessions (15-40 minutes each) per week, combined with 2 resistance training per week as well as motivational coaching via telephone Nutritional counseling
  Arms: Intervention

SUMMARY:
The aim of the study is to test the efficacy, feasibility, and safety of a bicycle exercise followed by an intensive lifestyle intervention for 3 months in patients with recent onset and medically untreated type 2 diabetes.

DETAILED DESCRIPTION:
Lifestyle intervention is a fundamental aspect in the treatment of type 2 diabetes. Implementation of lifestyle changes early after diagnosis often suffices to control metabolic dysregulation and may even have a durable impact. However, implementation of these changes is often difficult for multiple reasons including noncompliance as well as doubt on efficacy of sport and diet changes compared to drugs. Furthermore, most patients with type 2 diabetes remain asymptomatic for a prolonged period of time. Thus, they lack an immediate relief of symptoms and do not feel the benefit of changes in lifestyle. Often, untreated type 2 diabetes first manifests itself with symptoms of polyuria and polydipsia. This offers a unique opportunity to demonstrate the potential of lifestyle changes. However, in daily practice, symptomatic patients with polyuria and polydipsia or with HbA1c levels >10% at diagnosis are typically referred to an emergency room, hospitalized and treated with drugs as a first line treatment.

In the present study, we aim to implement a lifestyle intervention as a first-line treatment in recent onset type 2 diabetes. In the emergency room, the bed will symbolically be removed and the patient requested to perform a bicycle exercise. Non-ER patients will be invited to perform the bicycle exercise as soon as possible. We expect from this educational trigger that patients will realize the therapeutic power of sport. Preliminary interventions using this approach at our emergency room demonstrated the potential of such an intervention. However, internal and external validation, efficacy and safety of a lifestyle intervention in an emergency room remain to be shown in a multi-center controlled study.

The primary endpoint of this study is achievement of metabolic control without anti-diabetic medication 3 months after study enrollment. For the purpose of this study, metabolic control is defined as an HbA1c below a target stratified for three groups according to HbA1c at baseline: HbA1c >14% a target of < 10%; HbA1c < 14% and > 10% a target of < 8%; HbA1c < 10% a target of < 7.5%.

Patients will be randomized either to standard care or to a bicycle exercise followed by an intensive lifestyle intervention on top of non-pharmacological standard care.

After rehydration, patients allocated to the intensified lifestyle intervention group will be instructed to perform 30 minutes of bicycle exercise at 60 % of the calculated maximum heart rate (according to Franckowiak et al.) followed by an intensive lifestyle intervention. Patients will be discharged if the clinical status is stable and no comorbidities require further hospitalization. Follow-up visits at the Clinic of Endocrinology for further instructions and consultation will be carried out after 2, 7, 30, 60 and 90 days, half a year and a year.

In order to monitor blood glucose levels, patients will be instructed on visit 2 to take measurements at home and will be asked to send their fasting glucose levels of the first week to the study team for monitoring of the metabolic situation. This will also be done in the week before visits of day 30 and 90.

The schedule for the intervention arm consists of 3 to 5 aerobic training sessions (duration 15-40 minutes each) and 2 resistance trainings per week, as well as weekly motivational coaching via telephone by the study psychologist. Everyday activity will be objectively monitored using the patient's mobile phone and a blinded actigraph (activity tracker). Exercise sessions will be monitored by weekly phone calls and documented. To assess baseline physical activity all patients will fill in the SIMPAQ questionnaire at baseline and at 6 months.

Measurement of clinical parameters (heart rate, blood pressure), venous blood gas analysis (pH, pCO2, base excess, bicarbonate) at baseline and 120 min after beginning of bicycle exercise. Blood glucose levels at baseline and 30, 60 and 120 min after beginning of bicycle exercise. Blood glucose levels, vital parameters, concomitant medication after 2, 7, 30, 60 and 90 days; HbA1c at baseline, 2 (only intervention group), 3 and 6 months and one year; physical activity at baseline, 3 and 6 months. In the intervention group additional self-measurements of blood glucose levels during the first week and within the week before visit at day 30 and 90 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Type 2 diabetes diagnosed within the last two years according to the American Diabetes Association (ADA) criteria
* Age ≥ 18 years
* HbA1c ≥ 7.5 %

Exclusion Criteria:

* Clinically instable patient as defined by the physicians on duty including signs of new cardiac ischemia in the ECG, systolic blood pressure ≥ 200 mmHg, fever ≥ 38.5 °C, symptoms of SIRS or reduced vigilance.
* Anti-diabetic medication for ≥ 24 hours
* Inability to perform a bicycle exercise during 30 minutes
* Previous lifestyle-intervention by an endocrinologist
* Engagement in physical activity more than five times per week
* Enrollment in other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
metabolic control | 3 months
  fasting glucose < 7.6 mM and HbA1c below a target stratified for three groups according to HbA1c at baseline.

SECONDARY OUTCOMES:
Absolute HbA1c reduction per stratification group | 3 months
  Absolute HbA1c (% points) reduction after 3 months per stratification group (groups consist of HbA1c >14%; HbA1c <14% and >10%; HbA1c <10%)
Absolute HbA1c reduction per stratification group | 6 months
  Absolute HbA1c (% points) reduction after 6 months per stratification group (groups consist of HbA1c >14%; HbA1c <14% and >10%; HbA1c <10%)
Proportion of patients achieving HbA1c target in each stratification group | 3 months
  Proportion (%) of patients achieving target per stratified group after 3 months without anti-diabetic medication other than Metformin (groups consist of HbA1c >14%, HbA1c <14% and >10% and HbA1c <10%)
Feasibility of bicycle exercise at study enrollment in the ER | 2 hours
  Feasibility of bicycle exercise at study enrollment in the ER, defined as absence of problem reports through the study team
Proportion of patients achieving HbA1c target in each stratification group | 6 months
  Proportion (%) of patients achieving target per stratified group after 6 months without anti-diabetic medication other than Metformin (groups consist of HbA1c >14%, HbA1c <14% and >10% and HbA1c <10%)
Changes in heart rate after bicycle intervention | 2 hours
  Changes in heart rate (beats per minute) at the end and 120 min after bicycle exercise in the emergency room compared to baseline
Changes in respiratory rate after bicycle intervention | 2 hours
  Changes in respiratory rate (breaths per minute) at the end and 120 min after bicycle exercise in the emergency room compared to baseline
Changes in blood pressure after bicycle intervention | 2 hours
  Changes in blood pressure (mmHg) at the end and 120 min after bicycle exercise in the emergency room compared to baseline
Changes in blood glucose after bicycle intervention | 2 hours
  Changes in blood glucose (mmol/l) at the end and 120 min after bicycle exercise in the emergency room compared to baseline
Changes in pH after bicycle intervention | 2 hours
  Changes in pH at the end and 120 min after bicycle exercise in the emergency room compared to baseline
Changes in base excess after bicycle intervention | 2 hours
  Changes in base excess (BE) at the end and 120 min after bicycle exercise in the emergency room compared to baseline
Changes in bicarbonate after bicycle intervention | 2 hours
  Changes in bicarbonate (mmol/l) at the end and 120 min after bicycle exercise in the emergency room compared to baseline
Incidence of exercise related Adverse Events (Safety) during bicycle exercise in the ER | 2 hours
  Incidence of exercise related Adverse Events (cardiac, circulatory, pulmonary, neurologic complications) during bicycle exercise after diabetes diagnosis in the ER
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 6 months
  Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) during intensive lifestyle intervention after new diagnosis of type 2 diabetes
Re-hospitalization rate | 3 months
  Re-hospitalizations within 3 months after discharge from the emergency room.
Re-consultation rate | 3 months
  Rate of unplanned re-consultations within 3 months after discharge from the emergency room.
Changes in HbA1c at 6 months | 6 months
  Changes in HbA1c (in % points) at 6 months compared to baseline assessed by blood sample
Changes in physical activity at 6 months | 6 months
  Changes in physical activity at 6 months compared to baseline assessed by SIMPAQ questionnaire and actigraph.
  The SIMPAQ (Simple Physical Activity Questionnaire) measures daily physical activity. Time spent sedentary and active is measured in hours per day.
Number of antidiabetic medication at 30 days | 30 days
  Number of antidiabetic medication at 30 compared to baseline in both arms
Number of antidiabetic medication 60 days | 60 days
  Number of antidiabetic medication 60 days compared to baseline in both arms
Number of antidiabetic medication at 90 days | 90 months
  Number of antidiabetic medication at 90 days compared to baseline in both arms
Dosage of antidiabetic medication at 30 | 30 days
  Dosage of antidiabetic medication at 30 days compared to baseline in both arms
Dosage of antidiabetic medication at 60 days | 60 days
  Dosage of antidiabetic medication at 60 days compared to baseline in both arms
Dosage of antidiabetic medication at 90 days | 90 days
  Dosage of antidiabetic medication at 90 days compared to baseline in both arms
Quality of life by SF-36 Questionnaire | 6 months
  Quality of life at 6 months in intervention group as compared to standard of care as assessed by SF-36 questionnaire. The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (3):
- Switzerland (3):
  - University of Basel, Basel, Canton of Basel-City
  - Cantonal Hospital Olten, Olten, Canton of Solothurn
  - Hopital du Jura, Delémont

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT03827382/Prot_001.pdf